CLINICAL TRIAL: NCT04966143
Title: A Study of CLDN18.2 Chimeric Antigen Receptor T Cells in the Treatment of Advanced Pancreatic Cancer
Brief Title: Clinical Study of LY011 in the Treatment of Advanced Pancreatic Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Longyao Biotechnology Inc., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY011C1001
Record Dates: First submitted 2021-07-12; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Biological: LY011

INTERVENTIONS:
Biological: LY011 — Targeting CLDN 18.2 Car-T injection

SUMMARY:
CLDN 18.2 chimeric antigen receptor T cells Clinical research plan for the treatment of recurrent or refractory pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* They were 18 to 70 years old, male or female;
* Definitive diagnosis is recurrent or refractory pancreatic cancer;
* Claudin 18.2 IHC staining was positive in tumor tissues;
* Life expectancy > 12 weeks;
* According to RECIST 1.1, there was at least one measurable tumor target;
* ECoG scores at screening, 24 hours before puncture and baseline (before treatment) were 0-1;
* Adequate organ function;
* Women of childbearing age with negative pregnancy test or male subjects must take effective and reliable contraceptive methods until 30 days after the end of treatment;
* Have enough understanding ability to voluntarily sign informed consent to participate in clinical research.

Exclusion Criteria:

* Pregnant or lactating women;
* HIV, syphilis spirochete or HCV serological positive;
* Any uncontrollable active infection, including but not limited to active tuberculosis, HBV infection (HBsAg positive, HBcAb positive, HBV DNA positive);
* The subjects were judged as clinically significant thyroid dysfunction by the investigators (serum thyroid hormone determination TT4, TT3, FT3, FT4, serum thyroid stimulating hormone TSH) and were not suitable to participate in this study;
* The side effects of the patients were not recovered to CTCAE ≤ 1;
* Subjects who are currently using steroids all over the body within 7 days before the pregnancy is taken out; Inhaled steroids are not excluded in the near future or in the near future;
* Previous allergies to immunotherapy and related drugs, severe allergies or allergies;
* T cells (including car-t, tcr-t) that have been modified by chimeric antigen receptor have been reported.
* The subjects had untreated or symptomatic brain metastasis;
* The subjects had heart disease which needed treatment or after treatment, hypertension was out of control (blood pressure > 160 mmHg / 100 mmHg);
* Subjects with or waiting for organ transplantation history;
* No other serious disease may limit subjects' participation in this trial
* The researchers assessed that subjects were unable or unwilling to comply with the requirements of the study program.
* It has abnormal signs of central nervous system diseases or abnormal results of nervous system detection, which has clinical significance;
* Subjects currently or had other malignant tumors that could not be cured within 3 years, except for in situ cervical or skin basal cell carcinoma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response rate（ORR） | 1month
  the proportion of patients with best overall response of complete response (CR) or partial response (PR), as per local investigator´s assessment and according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria

SECONDARY OUTCOMES:
Progression free survival（PFS） | 1 years
  Survival witouth observed progression at 2 years
Disease Control Rate（DCR） | 1 years
  DCR (CR+PR+SD) by RECIST v1.1
Duration of Response (DOR） | 1 years
  DOR was defined as the time from the first documented a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) to progressive disease (PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm.
Overal survival （OS） | 5 years
  survival at 5 years
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 1 year
  AEs according to CTCAE v 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China